CLINICAL TRIAL: NCT06911125
Title: Investigation of the Effects of Diadynamic Current and Transcutaneous Electrical Nerve Stimulation on Pain and Functionality in Individuals With Chronic Neck Pain
Brief Title: Electrical Stimulation in Individuals With Chronic Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Gülşen Taşkın, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KA23/207
Record Dates: First submitted 2025-03-12; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Pain; Neck Pain; Neck Pain Chronic; Pain Intensity Assessment; Functional Status
Keywords: Transcutaneous Electric Nerve Stimulation; Diadynamic Current; Neck pain Chronic
MeSH Terms: conditions — Pain; Neck Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENS (Experimental): While the results of the use of TENS, an electrotherapy method, in chronic neck pain are included in some studies, the evidence regarding the effects of diadynamic currents is quite limited.
  Interventions: Device: TENS
- Diadynamic Currents (Experimental): While the results of the use of TENS, an electrotherapy method, in chronic neck pain are included in some studies, the evidence regarding the effects of diadynamic currents is quite limited.
  Interventions: Device: Diadinamic Current

INTERVENTIONS:
Device: TENS — TENS will be applied paravertebrally using four electrodes in the neck and back areas. Self-adhesive electrodes specific to each participant will be used for the application. TENS will run on symmetrical biphasic current at 100 Hz and 120 microseconds. The current intensity is determined by the level at which the person perceives the current. The participants are informed that they will get a current, which may induce a pins-and-needles sensation. It is essential for them to perceive the current distinctly; the intensity should be sufficient to be sensed without causing discomfort. The duration of the treatment is 20 minutes. Participants will receive exercises to strengthen the muscles around the neck.
  All participants will receive treatment once a day, five days a week. A total of 15 sessions will be conducted over a duration of 3 weeks.
  Arms: TENS
Device: Diadinamic Current — Diadynamic current will be performed paravertebrally using two electrodes on the neck and back areas. Participant-specific self-adhesive electrodes will be utilized for the application. In diadynamic current, two distinct current modules, namely diphase-fixed (2 minutes) and short period (8 minutes), will be utilized. The cumulative duration of the treatment is 10 minutes. The program will provide the current intensity at the threshold perceived by the individual. The participants will be informed about the application as follows: 'You will receive a current; you may have a pins-and-needles sensation; it is crucial to perceive the current distinctly and thoroughly; the intensity should neither be insufficient to be felt nor excessive to cause discomfort.' Participants will receive exercises to strengthen the muscles around the neck.All participants will receive treatment once a day, five days a week. A total of 15 sessions will be conducted over a duration of 3 weeks.
  Arms: Diadynamic Currents

SUMMARY:
The primary objective of the study was to evaluate the effects of diadynamic current and transcutaneous electrical nerve stimulation on pain and function in participants with chronic neck pain. The secondary objective of the research was to strengthen the neck muscles and enable participants with chronic neck pain to carry out everyday tasks on their own.

DETAILED DESCRIPTION:
Chronic neck pain is a common problem in individuals of all ages. Approximately two-thirds of individuals experience neck pain at least once in their lifetime. The methods used to treat non-specific neck pain are conservative-oriented, with medical treatment and physiotherapy being the first-line modalities. Electrotherapy tools like transcutaneous electrical stimulation (TENS), interferential current, diadynamic current, laser, and ultrasound are used to treat chronic neck pain. So are thermal modalities like hot packs, cold packs, hydrotherapy, and infrared; exercise therapies like neuromuscular control, diversified therapeutic exercises, range of motion (ROM) exercises, and strengthening exercises; and interventions like massage, mobilization-manipulation, and traction.

Methods that reduce pain and improve function are essential in treatment. Electrotherapy is a commonly used treatment among physical therapy modalities. While the results of the use of TENS, an electrotherapy method, in chronic neck pain are included in some studies, the evidence regarding the effects of diadynamic currents is quite limited. The primary objective of the study was to evaluate the effects of diadynamic current and transcutaneous electrical nerve stimulation on pain and function in participants with chronic neck pain. The secondary objective of the research was to strengthen the neck muscles and enable participants with chronic neck pain to carry out everyday tasks on their own.

The study's hypotheses are as follows:

Hypothesis 1: There is a difference between the effects of diadynamic current and transcutaneous electrical nerve stimulation on pain in participants with chronic neck pain.

Hypothesis 2: There is a difference between the effects of diadynamic current and transcutaneous electrical nerve stimulation on functionality in participants with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

Participants must be aged 18 to 60. Participants must report chronic neck pain for a minimum duration of three months.

Participants experiencing pain must have a Visual Analog Scale (VAS) score of at least 3.

Exclusion Criteria:

Participants with a history of neck or shoulder surgery Participants diagnosed with a rheumatic or neurological disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain intensity change in participants with chronic neck pain. | The first evaluation will be done before the treatment, the treatment program will be applied for 3 weeks and the same evaluations will be done again after the treatment is over
  Visual Analog Scale will be used to assess pain intensity.
  Visual Analog Scale Participants will be instructed to indicate their average pain intensity during rest, activity, and sleep on a 10-centimeter (cm) line, where 0 represents no pain and 10 represents horrible pain. The distance from the origin to the participant-marked point will be measured using a ruler, and pre-treatment pain scores will be recorded.

SECONDARY OUTCOMES:
Evaluation of functionality in participants with chronic neck pain. | The first evaluation will be done before the treatment, the treatment program will be applied for 3 weeks and the same evaluations will be done again after the treatment is over
  The Neck Disability Index is a scale that shows the functional status of the participants. The Neck Disability Index consists of ten questions related to pain intensity, personal care, lifting, reading, concentration, headaches, working, driving, sleeping, and recreational activities. For each question, there are 6 options ranging from 0 to 5 points. The questionnaire is evaluated out of a maximum of 50 points. "0 points" means no restrictions; "50 points' means full disability. "0-4 points" means no restriction, "5-14 points' means slightly restricted, "14-24 points' means moderately restricted, "25-34 points' means severely restricted, and "35 and above' means completely restricted.

OTHER OUTCOMES:
Overall pain | The first evaluation will be done before the treatment, the treatment program will be applied for 3 weeks and the same evaluations will be done again after the treatment is over
  McGill Pain Questionnaire- Short Form will be used to assess the overall pain of participants.
  McGill Pain Questionnaire- Short Form The McGill Pain Questionnaire Short Form is sufficiently sensitive to determine the efficacy of treatment interventions in alleviating pain. The questionnaire comprises 15 characteristics evaluated on a 4-point scale (the initial 11 evaluate the kind of pain, while the final 4 measure the emotional dimension): 0 = none, 1 = mild, 2 = moderate, 3 = severe.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşen Taşkın, Assist. Prof., Study Director — Afyonkarahisar Health Science University
Locations (1):
- Afyonkarahisar Health Science University, Türkiye, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No